CLINICAL TRIAL: NCT04006418
Title: A Registered Cohort Study on Spastic Paraplegia
Status: Recruiting | Type: Observational
Sponsor: Wan-Jin Chen (Other)
Responsible Party: Sponsor-Investigator, Wan-Jin Chen, The Vice-Director for the Department of Neurology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH OF FMU[2019]194
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Spastic Paraplegia
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Hereditary Spastic Paraplegias(HSP) and related disorders in a prospective multicenter natural history study, to assess the clinical, genetic and epigenetic features of patients with Spastic Paraplegias to optimize clinicalmanagement..

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of spastic paraplegia
* Clinical diagnosis of patients with spastic paraplegia
* Unrelated healthy controls

Exclusion Criteria:

* Decline to participate.
* There are serious interferences with individual participation and adherence to the research protocol, including but not limited to neurological, psychological, and/or medical conditions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed in hosipital and their's family
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2039-12 (Estimated); Study Completion 2049-12 (Estimated)

PRIMARY OUTCOMES:
Spastic Paraplegia Rating Scale (SPRS) | 6 months
  Disease severity will be assessed by application of the Spastic Paraplegia Rating Scale (SPRS), a clinical rating scale measuring disease severity in Hereditary Spastic Paraplegia (Schule et al. Neurology 2006). The SPRS contains 13 items, each ranging from 0 to 4 points. The total score is calculated as the sum of all items, yielding a range for the total score between 0 and 52. Hereby, higher SPRS total scores indicate more severe disease.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital Fujian Medical University, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang F, Hu J, Xiao Z, Lin C, Huang Z, Wang N, Liu Y. Spinal cord cross sign: a potential marker for hereditary spastic paraplegia type 5. Neuroradiology. 2025 Apr;67(4):1081-1090. doi: 10.1007/s00234-025-03543-y. Epub 2025 Jan 24. PMID 39853345
- [Derived] Tu Y, Liu Y, Fan S, Weng J, Li M, Zhang F, Fu Y, Hu J. Relationship between brain white matter damage and grey matter atrophy in hereditary spastic paraplegia types 4 and 5. Eur J Neurol. 2024 Aug;31(8):e16310. doi: 10.1111/ene.16310. Epub 2024 Apr 23. PMID 38651515
- [Derived] Qiu YS, Zeng YH, Yuan RY, Ye ZX, Bi J, Lin XH, Chen YJ, Wang MW, Liu Y, Yao SB, Chen YK, Jiang JY, Lin Y, Lin X, Wang N, Fu Y, Chen WJ. Chinese patients with hereditary spastic paraplegias (HSPs): a protocol for a hospital-based cohort study. BMJ Open. 2022 Jan 11;12(1):e054011. doi: 10.1136/bmjopen-2021-054011. PMID 35017251
- [Derived] Lin Q, Liu Y, Ye Z, Hu J, Cai W, Weng Q, Chen WJ, Wang N, Cao D, Lin Y, Fu Y. Potential markers for sample size estimations in hereditary spastic paraplegia type 5. Orphanet J Rare Dis. 2021 Sep 19;16(1):391. doi: 10.1186/s13023-021-02014-w. PMID 34538260